CLINICAL TRIAL: NCT02910544
Title: The Association Between Weight Loss and Changes in Physical Activity in Overweight/Obese Individuals With Knee Osteoarthritis: An Observational Cohort Study
Brief Title: Weight Loss and Physical Activity in Overweight/Obese Individuals With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Parker Research Institute (Other)
Responsible Party: Principal Investigator, Henrik Gudbergsen, MD, PhD, Parker Research Institute
Other Study IDs: 137.01
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Intensive dietary intervention: Supervised dietary weight loss program lasting 8 weeks.
  Interventions: Dietary Supplement: Intensive dietary intervention

INTERVENTIONS:
Dietary Supplement: Intensive dietary intervention — Participants receive a hypo-caloric formula diet containing 800 to 1,000 kcal/day. The formula diet consists of ready-to-use meal bars and powders to mix with water to make shakes, soups, or porridge. The weight loss programme consists of an 8-week period with full meal replacement by a standard liquid energy intake protocol. To facilitate compliance with the programme, participants will be scheduled for weekly facility-based group sessions with 6-8 participants led by a dietician. The recommendations for daily nutrient intake will be met.

SUMMARY:
This is a substudy to a randomised trial investigating the effect of liraglutide on body weight and pain in overweight or obese patients with knee osteoarthritis (NCT02905864). In the parent trial, patients will be subjected to an 8-week diet intervention phase including a low-calorie diet and dietetic counselling, after which.they will be randomised to receive either liraglutide 3 mg or liraglutide 3 mg placebo as an add-on to dietetic guidance on re-introducing regular foods and a focus on continued motivation to engage in a healthy lifestyle.

This substudy aims to investigate any changes in physical activity associated with the initial 8-week weight loss intervention.

DETAILED DESCRIPTION:
The investigators aim to describe changes in physical activity associated with a significant weight loss among overweight/obese individuals with knee OA. The investigators will take advantage of the planned trial "Effect of liraglutide on body weight and pain in overweight patients with knee osteoarthritis: A randomised, double blind, placebo-controlled, parallel group, single-centre trial" (the parent trial) in which a significant weight loss is sought achieved over 8 weeks by means of intensive dietary counseling and meal replacement in overweight/obese individuals with knee OA.

The investigators hypothesize that weight loss is associated with a decrease in daily time spent physically inactive.

Physical activity is measured using accelerometer based recordings using a wearable sensor that continuously records physical activity over the entire weight loss program (8 weeks). The sensor is miniaturised, discretely worn on the thigh, and is waterproof. Thus the measurements interfere minimally with the participants daily life.

ELIGIBILITY:
Further Inclusion Criteria:

* Eligible for parent trial (NCT02905864)
* Owner of a smart phone

Exclusion Criteria:

* Known allergies against band-aids

The eligibility criteria for this sub-study (i.e. owner of a smartphone and no known allergies against Band-Aids) are not considered requirements for participation in the parent study. Nor will any violation of this sub-study protocol affect participation, care, or attention given from the parent study.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants eligible for parent trial (NCT02905864), i.e. overweight/obese individuals with knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in time spent inactive (minutes) | week -8 to week 0
  Physical activity is recorded using an accelerometer based system with a built in algorithm for detection of standardised activities. Inactivity is defined as activities done sitting or lying down.

CONTACTS AND LOCATIONS:
Locations (1):
- The Parker Institute, Frederiksberg, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided